CLINICAL TRIAL: NCT01393353
Title: A Computerized, Multidimensional and Disease Specific Training of Cognition in Patients With M. Parkinson
Brief Title: Cognitive Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHBS
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Mental Competence
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer game (Sham Comparator): Nintendo Wii
  Interventions: Other: computer game
- Cognitive Training with Cogniplus (Experimental): CogniPlus
  Interventions: Other: Cognitive Training

INTERVENTIONS:
Other: Cognitive Training
  Arms: Cognitive Training with Cogniplus
Other: computer game
  Arms: Computer game

SUMMARY:
The study evaluates a computerized cognitive therapy in patients with Parkinson's disease who have a mild cognitive impairment or mild dementia. The control group is "trained" using Nintendo Wii. The main outcome parameter is a neuropsychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease and mild cognitive impairment (MCI) or mild dementia

Exclusion Criteria:

* Moderate or severe dementia, other pathologies of the brain, physical conditions that prevent the participation, unsufficient knowledge of german, pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Neuropsychological parameters: Tests of episodic memory, working memory, executive functions, visio-construction | Neuropsychological assessment immediatly before and after the training and 6 month later
  Neuropsychological tests: mini mental status (MMS), Clock drawing test, Boston Naming Test, Calculating, Semantic Fluency, Phonematic Fluency, California Verbal Learning Test, Corsi Block Tapping Test, Trail Making Test, Digit Span, Testbatterie zur Aufmerksamkeitsprüfung (alteredness, Working Memory, Divided Attention, Flexibility), Wisconsin Card Sorting Test, Apraxias, 5 Points Test, Mosaik Test

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof., Principal Investigator — University Hospital Basel, Neurology
Locations (1):
- University Hospital Basel, Basel, Switzerland